CLINICAL TRIAL: NCT05687136
Title: A Molecularly Driven Phase 1b Dose Escalation and Dose Expansion Study of the DNA-PK Inhibitor Peposertib (M3814) in Combination With the ATR Inhibitor M1774
Brief Title: Testing the Combination of Two Anti-cancer Drugs, Peposertib (M3814) and Tuvusertib (M1774) for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-10210; NCI-2022-10210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10527 (Other: Dana-Farber - Harvard Cancer Center LAO); 10527 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2023-01-14; First posted 2023-01-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (peposertib, tuvusertib) (Experimental): Patients receive peposertib PO QD or BID daily on days 2-14 of cycle 1 and days 1-14 of subsequent cycles in combination with tuvusertib PO QD or BID daily on days 1-14 of each cycle. Cycles repeat every 28 days in the absence of disease progression, pregnancy, non-compliance, unacceptable toxicity, termination of the study or the study drug is no longer available. Patients also undergo tumor biopsy, blood sample collection, PET, CT, and MRI throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Peposertib; Procedure: Positron Emission Tomography; Drug: Tuvusertib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Tuvusertib — Given PO
  Other Names: ATR Kinase Inhibitor M1774; M 1774; M-1774; M1774

SUMMARY:
This phase I trial tests the safety, side effects and best dose of peposertib (M3814) in combination with tuvusertib (M1774) in treating patients with solid tumors that have spread to other places in the body (advanced). Peposertib and tuvusertib stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of peposertib (M3814) in combination with tuvusertib (M1774). (DOSE ESCALATION AND EXPANSION COHORT) II. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of the combination of peposertib (M3814) and tuvusertib (M1774). (DOSE ESCALATION COHORT)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the pharmacokinetic (PK) profiles of peposertib (M3814) and tuvusertib (M1774) when administered in combination.

EXPLORATORY OBJECTIVES:

I. To explore correlations between pharmacodynamic (PD) and predictive biomarkers (gammaH2AX, phospho-KAP1 and phospho-RPA) with clinical outcomes.

II. To explore correlations between baseline genomic alterations of ataxia-telangiectasia mutated (ATM) or markers of replicative stress, ATM expression by immunohistochemistry (IHC), RAD5' foci formation with clinical outcomes.

III. To determine metrics of anticancer activity including the objective response rate (ORR) and progression-free survival (PFS).

OUTLINE: This a dose-escalation study of peposertib and tuvusertib, followed by a dose-expansion study.

Patients receive peposertib orally (PO) once (QD) or twice (BID) daily on days 2-14 of cycle 1 and days 1-14 of subsequent cycles in combination with tuvusertib PO QD or BID daily on days 1-14 of each cycle. Cycles repeat every 28 days in the absence of disease progression, pregnancy, non-compliance, unacceptable toxicity, termination of the study or the study drug is no longer available. Patients also undergo tumor biopsy, blood sample collection, positron emission tomography (PET), computed tomography (CT), and magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up for a minimum of 30 days after removal from treatment or until initiating a new anticancer therapy or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* For the dose escalation and dose expansion phases, patients must have genomic (tumor next-generation sequencing [NGS], circulating tumor deoxyribonucleic acid [ctDNA], fluorescence in situ hybridization [FISH], etc.) or immunohistochemical evidence of inactivating ATM mutations, MYC amplification, mutation of FBXW7, CCNE1 amplification, SWI/SNF member mutation (ARID1A, PBRM1, SMARCA4, ARID2, ARID1b, SMARCB1, SMARCA2, SS18), and ATRX/DAXX. Mutations may be germline or somatic. All mutations/alterations must be approved by the overall principal investigator (PI). Other SWI/SNF mutations may be considered after discussion with the overall PI.
* Progression on at least one prior standard therapy.
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of peposertib (M3814) in combination with tuvusertib (M1774) in patients < 18 years of age, children are excluded from this study.
* Life expectancy > 3 months.
* Eastern cooperative oncology group (ECOG) performance status =< 2 (Karnofsky >= 60%).
* Measurable disease by response evaluation criteria in solid tumors (RECIST) 1.1 (RECIST) 1.1 non-measurable disease permitted for the dose escalation portion).
* Hemoglobin >= 9 g/dL.
* Absolute neutrophil count >= 1,500/mcL.
* Platelets >= 1000,000/mcL.
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 3 × institutional ULN or =< 5.0X the ULN if liver metastases are present.
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73m^2.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Anti-retroviral therapy agents must be considered for potential drug-drug interactions per exclusion.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Able to swallow whole capsules or tablets.
* Willing to undergo paired biopsies (expansion arm).
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  * Female patients of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 6 months after the last dose of study medication.
  * Male patients of reproductive potential must agree to avoid impregnating a partner while receiving study drug and for 3 months after the last dose of study drug by complying with adequate methods of contraception.
  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible.

Exclusion Criteria:

* Patients who have received immunotherapy within 21 days of Cycle 1 Day 1.
* Patients who have received therapeutic radiation therapy within 21 days, or palliative radiation therapy within 7 days, of Cycle 1 Day 1.
* Patients who have undergone major surgery within 21 days of Cycle 1 Day 1.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia, controlled endocrine toxicity (e.g., hypothyroidism), and cutaneous toxicity which will be permitted at Grade 2.
* Patients who are receiving any other investigational agents.
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate central nervous system (CNS) specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to peposertib (M3814) and tuvusertib (M1774).
* Patients who cannot discontinue concomitant medications or herbal supplements that are strong inhibitors or strong inducers of cytochrome P450 (CYP) isoenzymes, CYP1A2, CYP3A4/5, CYP2C19, and CYP2C9. Concomitant use of substrates hMATE1, hMATE2, and CYP3A4/5 substrates with a narrow therapeutic index are also excluded. Opioids may interact with these enzymes; use of opioids while on study is allowed but should be closely monitored. Concomitant administration of sensitive substrates of P-gp, BCRP, OCT1, OATP1B1, and OATP1B3 should be avoided (if the use is unavoidable, carefully monitor patients for signs of increased toxicity). Patients may confer with the study doctor to determine if alternative medications can be used. The following categories of medications and herbal supplements must be discontinued for at least the specified period of time before the patient can be treated:

  * Strong inducers of CYP1A2, CYP3A4/5, CYP2C19, and CYP2C9: >= 3 weeks prior to study treatment.
  * Strong inhibitors of CYP1A2, CYP3A4/5, CYP2C19, and CYP2C9: >= 1 week prior to study treatment.
  * Substrates of hMATE1, hMATE2, CYP3A4/5, P-gp, BCRP, OCT1, OATP1B1, and OATP1B3 with a narrow therapeutic index: >= 1 day prior to study treatment.
* Patients who cannot discontinue proton-pump inhibitors (PPIs). H-2-receptor antagonist should be held during the 2 weeks of concurrent dosing with peposertib (M3814). There is no H-2-receptor antagonist restriction during the off weeks without peposertib (M3814) dosing. H-2-receptor antagonists should not be taken within 12 hours before or 2 hours after tuvusertib (M1774). Antacids should not be taken within 2 hours before or 2 hours after tuvusertib (M1774).
* Patients who received hematopoietic growth factor (e.g., granulocyte colony-stimulating factor, erythropoietin) within 14 days prior to the first dose of study intervention.
* Patients with uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* QTcF (using the Fridericia correction calculation) of >= 470 msec
* Pregnant women and women who are breastfeeding are excluded from this study because the effects of the study drugs on the developing fetus are unknown.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as assessed by the treating investigator may be included with the approval of the sponsor-investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | Up to 28 days
Incidence of adverse events | Up to week 12
  Descriptive statistics will be used for safety in the Phase 1b escalation study. Patients will be included in this analysis if they receive at least one dose of any study treatment. For toxicity reporting, all adverse events will be graded and analyzed using Common Terminology Criteria for Adverse Events (CTCAE). Type of adverse events, intensity (grading), and attribution will be provided in a listing. All adverse events resulting in discontinuation, dose modification, and/or dosing interruption, and/or treatment delay of drug will also be summarized. Laboratory test results will be classified according to CTCAE.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) analysis | Pre, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hour (h) post dose on cycle (C)1 day (D)1, pre, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 h post dose on C1D10 (dose-escalation); pre, 0.5, 1,1.5, 2, and 3 h post dose on C1D1 and C1D10 (dose-expansion)
  Peposertib (M3814) and tuvusertib (M1774) concentrations in these samples will be quantitatively measured using a liquid chromatography/tandem mass spectrometric method. The individual PK parameters will be derived: maximum concentration (Cmax), time to maximum concentration (Tmax), are under the curve (AUC), half life (T1/2), apparent oral clearance (Cl/F), and apparent volume of distribution in steady state (Vss/F) using non-compartmental methods with the software WinNonlin, as feasible. Advanced population PK methods may be employed to assess the link between drug exposure and biological effects and efficacy. The PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) calculated for each dose level. PK parameters (e.g., T1/2, Cmax, Cl, and AUC) will be compared across dose level using nonparametric statistical testing techniques.

OTHER OUTCOMES:
Pharmacodynamics (PD) | After registration and before C1D1 and at C1D10
  Will be assessed using the changes in gammaH2AX, phosphorylated biomarkers (e.g., NBS1, RPA, KAP1), and gene expression by ribonucleic acid sequencing before and on treatment. Correlation between mutation status and immunohistochemistry results with ATM will be descriptive as well.
Overall response rate (ORR) | Up to 2 years
  In the phase 1b expansion, the ORR will be estimated by the proportion of patients who achieve complete or partial response as their best response to treatment. ORR will be accompanied by a 95% confidence interval estimated using exact binomial methods.
Progression free survival (PFS) | Up to 2 years
  The time to event endpoint PFS will be estimated with the Kaplan Meier methodology. Median and event-free rate at selected time points will be provided with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Cote, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (6):
- United States (6):
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm